CLINICAL TRIAL: NCT04686019
Title: "More Air - Better Performance - Faster Recovery": Study Protocol for a Randomised Controlled Trial of the Effect of Inspiratory Muscle Training for Adults Post-stroke
Brief Title: More Air - Better Performance - Faster Recovery
Acronym: IMT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Sygekassernes Helsefond (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-16-02-279-20
Record Dates: First submitted 2020-10-28; First posted 2020-12-28 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2020-10

CONDITIONS: Functional Independence; Respiratory Insufficiency
Keywords: Stroke,; Functioning; Fatigue; Voice volume
MeSH Terms: conditions — Respiratory Insufficiency; Stroke; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: External assessor unknown to the participants of the intervention group and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): * 2 x IMT (5-10 min) 2 times a day 7 days a week for 3 weeks with or without supervision
  * Log-book
  * Conventional neurorehabilitation
  Interventions: Other: Inspiratory muscle training (IMT)
- Control group (Active Comparator): Conventional neurorehabilitation
  Interventions: Other: Inspiratory muscle training (IMT)

INTERVENTIONS:
Other: Inspiratory muscle training (IMT) — IMT and conventional neurorehabilitation - treatment as usual. The intervention group will add-on IMT sessions exercising at 30 % of MIP. MIP is measured by instructing the patient to perform five forceful inspirations against an occluded mouthpiece (Power Breath). The best score is multiplied by 0.3 to determine the resistance. IMT is performed with IMT Threshold flute with the calculated resistance. During the measurement with Power Breath the patient sits straight up and uses nose clip. The patient can receive help to hold the Power Breath if necessary.
  One session of IMT with IMT threshold flute consists of 2 times 15 inspirations in normal breathing rhythm (5-10 min). Patients in the intervention group perform 2 sessions a day (morning and evening), training is performed prior to a meal, 7 days a week for 3 weeks.

SUMMARY:
The objective of this study is to investigate i) the effect of 3 weeks IMT to adults post-stroke to maximal inspiratory pressure (MIP) and ii) the effects of 3 weeks IMT to the degree of dependency in activities of daily living, endurance in gait, fatigue, voice volume, phonation endurance, and expiratory function.

Methods/Design: Randomised controlled trial (RCT) comparing IMT to conventional neurorehabilitation (usual practise). 80 patients, with reduced maximal inspiration pressure (MIP) hospitalized at a specialized neurorehabilitation hospital in Denmark will be included.

DETAILED DESCRIPTION:
Background: Stroke results in varying disabilities physical, cognitive, emotional and/or social both in short term and long term. Motor impairments are significantly persistent consequences post-stroke among these are decreased respiratory muscle function, decreased ability to expand thorax and postural dysfunction. These deficits influence the patient's ability in daily activities, fatigue, endurance and quality of life. Inspiratory muscle training (IMT) is training to improve the strength and endurance of diaphragm and the external intercostal muscles. The objective of this study is to investigate i) the effect of 3 weeks IMT to adults post-stroke to maximal inspiratory pressure (MIP) and ii) the effects of 3 weeks IMT to the degree of dependency in activities of daily living, endurance in gait, fatigue, voice volume, phonation endurance, and expiratory function.

Methods/Design: Randomised controlled trial (RCT) comparing IMT to conventional neurorehabilitation (usual practise). 80 patients, with reduced maximal inspiration pressure (MIP) hospitalized at a specialized neurorehabilitation hospital in Denmark will be included. The intervention group will add-on IMT sessions exercising at 30 % of MIP. Patients in the intervention group perform 2 sessions a day (One session of IMT with IMT threshold flute consists of 2 times 15 inspirations in normal breathing rhythm (5-10 min)), 7 days a week for 3 weeks. Training can be with or without supervision of physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* First time brain infarction or brain haemorrhage 0-6 month.
* Able to give written consent and being cognitive and communicative able to understand and participate in the maximal inspiration pressure test (MIP)
* Reduced MIP below gender and age specific normal standard

Exclusion Criteria:

* Diagnosis of myocardial infarction within the last 3 months
* Significant pulmonary disease (severe COPD), saturation below 90 if having COPD for others saturation below 92
* Neurological deficits other than stroke
* Facial palsy that affects proper labial occlusion
* Dizziness or nausea/vomiting during MIP-testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  Change of MIP assess with the Power Breath. This is an objective measurement to describe the inspiratory capacity. Age specific

SECONDARY OUTCOMES:
Functional Independence Measure (FIM) - both total score ( range from 18 to 126, with higher scores indicating more independence) and motor sub score (max 91) | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  to assess the degree of changed dependency in daily activities
Fatigue Severity Scale (FSS) | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  to measure change of fatigue (1-63) higher scores indicating more fatigue affected.
6-minutes walking test | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  to measure change of endurance
Voice volume | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  to measure change of voice volume by recording of an a-sound with the App Voice Analyst and to measure Phonation endurance (how long the a-sound last)
Expiratory function | Assessed 0-4 days before intervention, 0-4 days after ended intervention assessment and 3 months after ended intervention
  To measure change of Peak expiratory flow (PEF), Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC) and FEV1/FVC ratio will be assessed with a peak flow meter (Spirometry device Micro 6300)

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen F Nielsen, Professor, Study Chair — Hammel Neurorehabilitation and Research Centre, University of Aarhus, Hammel, Denmark
Locations (1):
- Regional Hospital Hammel Neurocenter, Hammel, Denmark

IPD SHARING:
Plan to Share IPD: No
no plan

REFERENCES:
- [Derived] Sorensen SL, Kjeldsen SS, Mortensen SS, Hansen UT, Hansen D, Pedersen AR, Pallesen H. "More air-better performance-faster recovery": study protocol for randomised controlled trial of the effect of post-stroke inspiratory muscle training for adults. Trials. 2021 Aug 28;22(1):575. doi: 10.1186/s13063-021-05551-8. PMID 34454573